CLINICAL TRIAL: NCT02404558
Title: An Open-label, Randomized, Parallel Group, Single-dose Study to Describe the Safety of IL-6 Receptor Blockade With Sarilumab or Tocilizumab Monotherapy in Japanese Patients With Rheumatoid Arthritis
Brief Title: Single-dose Study to Describe the Safety of Sarilumab and Tocilizumab in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDY14191; U1111-1163-1359 (Other: UTN)
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sarilumab (Experimental): Single subcutaneous (SC) dose of sarilumab
  Interventions: Drug: sarilumab SAR153191 (REGN88)
- Tocilizumab (Active Comparator): Single SC dose of tocilizumab
  Interventions: Drug: tocilizumab

INTERVENTIONS:
Drug: sarilumab SAR153191 (REGN88) — Pharmaceutical form:solution Route of administration: Subcutaneous injection
  Arms: Sarilumab
Drug: tocilizumab — Pharmaceutical form:solution Route of administration: Subcutaneous injection
  Arms: Tocilizumab

SUMMARY:
Primary Objective:

To describe the safety and tolerability, including laboratory abnormalities following a single dose of sarilumab or tocilizumab administered subcutaneously (SC) as monotherapy in Japanese patients with rheumatoid arthritis (RA).

Secondary Objectives:

To describe the laboratory abnormalities (absolute neutrophil count [ANC], platelet counts, total cholesterol, high-density lipoprotein [HDL] cholesterol, low-density lipoprotein [LDL] cholesterol, and liver function tests [LFTs]) following a single dose of sarilumab or tocilizumab administered SC as monotherapy in Japanese patients with RA.

To describe the pharmacokinetics (PK) of sarilumab and tocilizumab.

DETAILED DESCRIPTION:
Total study duration (per patient) is expected to be up to 71 days including screening (3 to 28 days before dosing).

ELIGIBILITY:
Inclusion criteria:

* Patients with rheumatoid arthritis (RA) as defined by the American College of Rheumatology (ACR)/European League against Rheumatism (EULAR) 2010
* Rheumatoid Arthritis Classification Criteria.
* ACR Class I-III functional status, based on the 1991 revised criteria.

Exclusion criteria:

* Patients less than 20 years of age.
* Prior treatment with any biologic anti-interleukin-6 (anti-IL-6) or interleukin-6 receptor (IL-6R) antagonist.
* Any parenteral or intraarticular glucocorticoid injection within 4 weeks prior to randomization.
* Treatment with prednisone higher than 10 mg or equivalent per day, or change in dosage within 4 weeks prior to randomization.
* Treatment with disease-modifying antirheumatic drugs (DMARDs), immunosuppressive agents, tumor necrosis factor (TNF) antagonists or any other RA-directed biologic agents within a certain amount of time prior to randomization.
* Participation in any clinical research study that evaluated an investigational drug or therapy within 5 half-lives or 60 days of the screening visit, whichever is longer.
* Active or suspected tuberculosis (TB) or at high risk of contracting TB.
* Fever, or chronic, persistent, or recurring infection(s) requiring active treatment.
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with adverse events | 6 weeks
Percentage of patients with potentially clinically significant laboratory abnormalities | 6 weeks
Change from baseline in laboratory parameters (hematology and biochemistry) | Baseline, Day 15
Weighted average of change from baseline in laboratory parameters (hematology and biochemistry) | Baseline, Day 15

SECONDARY OUTCOMES:
Assessment of PK parameter: maximum concentration (Cmax) | Day 1 to Day 43
Assessment of PK parameter: time to Cmax (tmax) | Day 1 to Day 43
Assessment of PK parameter: area under the curve from zero time until the last measurable concentration (AUClast) | Day 1 to Day 43
Change from baseline in laboratory parameters (hematology and biochemistry) | Baseline, Day 29 and Day 43
Weighted average of change from baseline in laboratory parameters (hematology and biochemistry) | Baseline, Day 29 and Day 43

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Japan (3):
  - Investigational Site Number 392001, Sendai
  - Investigational Site Number 392002, Sendai
  - Investigational Site Number 392003, Sendai

REFERENCES:
- [Derived] Kovalenko P, Paccaly A, Boyapati A, Xu C, St John G, Nivens MC, Davis JD, Rippley R, DiCioccio AT. Population Pharmacodynamic Model of Neutrophil Margination and Tolerance to Describe Effect of Sarilumab on Absolute Neutrophil Count in Patients with Rheumatoid Arthritis. CPT Pharmacometrics Syst Pharmacol. 2020 Jul;9(7):405-416. doi: 10.1002/psp4.12534. Epub 2020 Jun 20. PMID 32453485